CLINICAL TRIAL: NCT00395122
Title: Evaluation of the Diagnostic Ability of Optical Coherence Tomography With a Normative Database to Detect Band Atrophy of the Optic Nerve
Brief Title: Optical Coherence Tomography Measurements in Eyes With Band Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCT in band atrophy; FAPESP grant No 05/55326-1
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-11

CONDITIONS: Vision Disorders
Keywords: Band Atrophy; Optical Coherence Tomography; Scanning Laser Polarimetry; Chiasmal Lesions
MeSH Terms: conditions — Vision Disorders

INTERVENTIONS:
Device: Retinal nerve fiber layer and macular thickness measurements

SUMMARY:
The study is designed to evaluate the ability of optical coherence tomography and VCC scanning laser polarimetry to measure and identify the pattern of band atrophy of the optic nerve in patients with long standing chiasmal lesions. The hypothesis is that these new technologies are able to identify such pattern. The idea is that by using eyes with band atrophy one is able to investigate the ability of the new technologies in measuring the retinal nerve fiber layer particularly in the nasal and temporal portions of the optic nerve.

ELIGIBILITY:
Inclusion Criteria:Patients with long standing chiasmal lesions and temporal visual field defect with the following criteria:

1. Visual acuity better than 20/30
2. Refractive error less 5 spherical diopter and 3 cylinder diopter
3. Temporal field defect

Exclusion Criteria:

1. Presence of glaucoma and optic nerve anomalies
2. Anormal nasal field

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2006-10

PRIMARY OUTCOMES:
Retina nerve fiber layer measurements
Macular thickness measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mário LR Monteiro, MD, PhD, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Derived] Moura FC, Costa-Cunha LV, Malta RF, Monteiro ML. Relationship between visual field sensitivity loss and quadrantic macular thickness measured with Stratus-Optical coherence tomography in patients with chiasmal syndrome. Arq Bras Oftalmol. 2010 Sep-Oct;73(5):409-13. doi: 10.1590/s0004-27492010000500004. PMID 21225123